CLINICAL TRIAL: NCT05100329
Title: Safety, Tolerability, and Efficacy of Mitoxantrone Hydrochloride Liposome Injection in Patients With Advanced Pancreatic Cancer: A Multicenter, Open-label, Phase Ⅱ Study
Brief Title: A Study of Mitoxantrone Hydrochloride Liposome Injection in Patients With Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-026
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-06

CONDITIONS: Advanced Pancreatic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome Injection (Experimental): Patients will receive mitoxantrone hydrochloride liposome injection every 3 weeks (q3w, a cycle).
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome injection

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome injection — 20 mg/m^2, IV, on day 1 of every 3 weeks (q3w, a cycle)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of mitoxantrone hydrochloride liposome injection in patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase Ⅱ study aimed to evaluate the safety, tolerability, and efficacy of mitoxantrone hydrochloride liposome injection in patients with advanced pancreatic cancer. Patients enrolled in this study will receive mitoxantrone hydrochloride liposome injection every 3 weeks (q3w, a cycle) until disease progression, intolerable toxicity, death, or withdrawal by investigator or patient decision (a maximum of 8 cycles).

ELIGIBILITY:
Inclusion Criteria:

1. Patients fully understand and voluntarily participate in this study and sign informed consent;
2. Aged 18-75 years (inclusive), without gender limitation;
3. Histologically or cytologically confirmed advanced pancreatic tumors;
4. Patients with locally progressive or metastatic pancreatic cancer who have disease progression after receiving first line or above standard treatment.
5. At least one measurable lesion according to RECIST v1.1 at baseline;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2;
7. Adequate organ function defined as (No G-CSF treatment or blood transfusion within 2 weeks prior to the first dose):

   * Absolute neutrophil count (ANC) ≥1.5*10^9/L;
   * Hemoglobin ≥ 90 g/L;
   * Platelet count ≥ 100 * 10^9/L;
   * Creatinine ≤1.5 * upper limit of normal (ULN);
   * Total bilirubin ≤2 * ULN;
   * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 3 * ULN (≤ 5 * ULN in patients with hepatic metastasis);
   * Coagulation: prothrombin time (PT) or International Normalization Ratio (INR) ≤1.5 * ULN.
8. Female patients must have a urine or blood HCG negative test before enrolment (except for menopause and hysterectomy); Patients and their partners must agree to use effective contraceptive measures during the study until 6 months after the end of the last dose.
9. Good compliance and willingness to cooperate with follow-up visits.

Exclusion Criteria:

1. History of severe allergy to mitoxantrone hydrochloride or any excipients of the study drug;
2. History of other malignant tumor in previous 3 years, not including cured cervical carcinoma in situ, skin basal cell carcinoma or squamous cell carcinoma.
3. Cerebral or meningeal metastases;
4. Patients with chronic hepatitis B (HBsAg positive with HBV DNA ≥ 2000 IU/mL), chronic hepatitis C (HCV antibody positive with HCV RNA above the lower limit of detection of the study center), or human immunodeficiency virus (HIV) antibody positive;
5. Life expectancy < 3 months;
6. Previous treatment with adriamycin or other anthracyclines, with the total cumulative dose (doxorubicin equivalent) >350 mg/m^2;
7. AEs from the previous treatment have not resolved to ≤ Grade 1 based on CTCAE (except for the toxicity without safety risk judged by the investigator, such as alopecia, hyperpigmentation);
8. Patients with the following cardiac function defects:

   * Long QTc syndrome or QTc interval > 480 ms;
   * Complete left bundle branch block, II-III degree atrioventricular block;
   * Severe, uncontrolled arrhythmias requiring pharmacological treatment;
   * History of chronic congestive heart failure, NYHA ≥ grade 3;
   * Cardiac ejection fraction < 50% within 6 months prior to screening;
   * Heart valve disease with CTCAE ≥ grade 3;
   * History of myocardial infarction, unstable angina, severe ventricular arrhythmias, severe pericardial disease, or ECG evidence of acute ischemic or active conduction system abnormalities within 6 months prior to screening;
9. Uncontrollable hypertension (defined as a measured systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg under pharmacological control);
10. Malignant serous cavity effusion (e.g. pleural effusion, pericardial effusion, ascites);
11. Active bacterial, fungal or viral infections requiring intravenous infusion treatment within 1 week prior to the first dose;
12. Any anticancer treatment within 4 weeks prior to the first dose (e.g., radiotherapy, targeted therapy, immunotherapy, endocrine therapy, etc.); Traditional Chinese medicine or proprietary Chinese medicine with an approved oncology indication within 2 weeks prior to the first dose;
13. Enrolled in any other clinical trials within 4 weeks prior to the first dose;
14. Patients underwent major surgery within 12 weeks prior to the first dose, or have a surgical schedule during the study period;
15. Having a schedule of other anti-cancer treatment during the study period.
16. Deep vein thrombosis or arterial embolism within the previous 6 months, including but not limited to superior/inferior vena cava thrombosis, lower limb deep vein thrombosis, pulmonary embolism;
17. Lactating female;
18. Serious and/or uncontrolled medical condition that, in the judgment of the investigator, may affect the patient's participation in this study (including, but not limited to: diabetes not effectively controlled, kidney disease requiring dialysis, severe liver disease, life-threatening autoimmune and bleeding disorders, neurological disorders, etc.);
19. Not suitable for this study as decided by the investigator due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 3 years
  ORR is defined as the proportion of patients who have a best overall response of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 3 years
  OS is defined as the time from the date of first dose until the date of death from any cause.
Progression-free survival (PFS) | Up to approximately 3 years
  PFS is defined as the time from the date of first dose until the date of first documented progressive disease (PD) as per RECIST 1.1 or death from any cause, whichever occurs first
Disease control rate (DCR) | Up to approximately 3 years
  DCR is defined as the proportion of patients who have a response of CR/PR or stable disease (SD) as per RECIST 1.1.
Duration of response (DoR) | Up to approximately 3 years
  DoR is defined as the time from the first assessment of CR or PR until the date of first occurrence of progressive disease （PD） as per RECIST 1.1 or death from any cause, whichever occurs first.
Treatment-emergent adverse events (TEAEs) | Up to approximately 3 years

IPD SHARING:
Plan to Share IPD: No